CLINICAL TRIAL: NCT07150026
Title: An Exploratory Evaluation of the Safety and Efficacy of Vorinostat in Pitt Hopkins Syndrome Using an "N of 1" Study Design
Brief Title: An Exploratory Evaluation of the Safety and Efficacy of Vorinostat in Pitt Hopkins Syndrome
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Unravel Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RVL-001 Study 003; 20251103997 (Other: Instituto Nacional de Vigilancia de Medicamentos y Alimentos)
Record Dates: First submitted 2025-08-14; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pitt Hopkins Syndrome
Keywords: Pitt Hopkins; n of 1; interventional
MeSH Terms: conditions — Pitt-Hopkins syndrome | interventions — Vorinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose interventional arm (Experimental): vorinostat low dose 80mg/m2/day
  Interventions: Drug: Vorinostat (SAHA)
- High dose interventional arm (Experimental): vorinostat 160mg/m2/day dose
  Interventions: Drug: Vorinostat (SAHA)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vorinostat (SAHA) — oral suspension
  Other Names: suberoylanilide hydroxamic acid
  Arms: High dose interventional arm; Low dose interventional arm
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The study is an exploratory evaluation of the safety and efficacy of vorinostat in Pitt Hopkins syndrome. Each patient will be self-controlled in an adapted N-of-1 study design methodology with three treatment arms, including a 4-week placebo phase and two vorinostat dose arms, including every 8 weeks of daily dosing at a low dose of 80mg/m2/day and 8 weeks of a higher dose at 160mg/m2/day.

Key objectives of the study include:

* To confirm the safety and tolerability of oral vorinostat 80mg/m2/day and 160mg/ m2/day dose levels when administered to PTHS patients
* To identify the nature and magnitude of treatment response to vorinostat, as measured by changes in clinical and laboratory parameters indicative of trend towards benefit, as well as changes in mRNA expression (transcriptome response)
* Provide a data-driven justification for future study design and statistical analysis plan for subsequent clinical studies assessing safety and efficacy of vorinostat in PTHS

DETAILED DESCRIPTION:
Unravel Biosciences, Inc. ("Unravel") proposes to develop an orally administered, once daily novel treatment for the orphan drug indication of Pitt Hopkins syndrome. Unravel has utilized its proprietary drug discovery platform to identify drugs having potential therapeutic value for neurodevelopmental disorders caused by gene mutations shown to have a cascading effect on other genes. Unravel's platform combines human gene regulatory network-based computational drug prediction with in vivo screening in a population-level diversity, CRISPR-edited, Xenopus laevis tadpole disease model. Through use of Unravel's platform, the drug vorinostat ranked highly in predictive scoring for Pitt Hopkins syndrome. In work done for Rett syndrome, another orphan CNS disease with many molecular and phenotypic similarities to Pitt Hopkins syndrome, vorinostat broadly improved both CNS and non-CNS (e.g., gastrointestinal, respiratory, inflammatory) abnormalities in a pre-clinical mouse model of Rett syndrome. Vorinostat was the first treatment to demonstrate nonclinical efficacy across multiple organ systems when dosed after the onset of symptoms, and network analysis revealed a putative therapeutic mechanism for its cross-organ normalizing effects based on its impact on acetylation metabolism and post-translational modifications of microtubules, leading to the selection of vorinostat as a target candidate for further assessment in both Rett and Pitt Hopkins syndromes. The main hypotheses informing the goals and design of the study are as follows:

* Vorinostat is safe and tolerable when dosed in typical Rett patients at dose levels up to 160mg/m2/day
* At a molecular level, vorinostat mitigates the impact of the underlying TCF4 gene mutation in PTHS patients by restoring downstream mRNA synthesis, as measured by transcriptome data
* Vorinostat provides clinical benefit to Pitt Hopkins patients by reducing frequency and severity of clinical signs/symptoms and improving patient quality of life

The study is designed as an exploratory, proof of concept trial to investigate the study hypotheses as stated above and to achieve the primary goals of the trial. The study design adapts the well-known "n of 1" crossover study methodology (Guyatt, et.al., 1990, Kravitz, et.al., 2014), where each patient serves as their own control during comparative analyses of safety and efficacy. Up to 5 patients will be enrolled in the study to explore the hypothesis that vorinostat is a safe and potentially effective treatment for Pitt Hopkins syndrome. Each patient enrolled in the study will be exposed to a 4-week placebo study phase to generate baseline data that will serve as a control as well as two active drug phases with vorinostat treatment, starting at 80mg/m2/day dosing for 8 weeks, followed by dose escalation to 160mg/m2/day for 8 weeks. The study is designed to be single-blinded, where patients and their caregivers will not be aware of their treatment assignment in an attempt to minimize bias where practically possible, especially given the subjective nature of several of the endpoints being evaluated. Investigator, study staff, and sponsor will not be blinded to study treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥3 years of age and ≤ 21 years of age at time of screening
2. Clinical diagnosis of PTHS with documented pathologic mutation in the TCF4 gene
3. At time of screening, is in a post-regression phase with no degradation of ambulation, hand function, speech or communication skills in the 4 months prior to screening
4. Has been on a stable regimen of medication or non-pharmacological treatment for at least 4 weeks prior to the baseline visit
5. Has had a stable pattern of seizure activity for 4 weeks before screening
6. Can swallow medication or can take it by gastrostomy tube
7. Can wear actigraphy data logging device on wrist or ankle
8. If of childbearing potential, must agree to use a highly effective method of contraception during the study and for 3 months after the last study drug administration (i.e., abstinence from sexual activity, hormonal contraceptives associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system)
9. Subjects or their legally authorized representative must be able to provide an informed consent and have sufficient language skill to complete caregiver assessments in the language in which the study assessments are provided

Exclusion Criteria:

1. Has another clinically significant medical condition other than those related to their TCF4 mutation (e.g. diabetes mellitus, cardiovascular disease, renal disease, respiratory disease, hematological abnormalities, malignancy)
2. Has major surgery planned during the study period
3. Pregnant or nursing women
4. Has a history of brain injury, stroke, other cerebrovascular disease or hypoxic-ischemic encephalopathy
5. Has clinically significant abnormal vital signs at screening or baseline
6. Has an abnormal ECG at screening, including clinically significant QT prolongation
7. Has a clinically significant abnormal laboratory value at screening
8. Liver disease or transaminase levels > 1.5 times the upper limit of the normal range as determined during screening
9. Has a history of malignancy of any organ system within the past 5 years before screening
10. Is participating in or has participated in another clinical trial within 30 days prior to the screening visit
11. Has been treated with growth hormone, IGF-1, or insulin within 12 weeks of baseline
12. Is taking anticoagulant therapy or other HDAC inhibitors
13. Has had any change to their medication or non-pharmacological treatment within 4 weeks prior to the baseline visit
14. Life expectancy of less than 12 months.
15. Has a history of alcoholism or drug/chemical abuse within 2 years before screening.
16. In the investigator's opinion, is inappropriate for this study for any reason

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment-related adverse events | 20 weeks
  Treatment-related adverse events coded by MedDRA will be compared qualitatively between low dose treatment, high dose treatment, and placebo groups
Drug tolerability as measured by number of treatment discontinuations | 20 weeks
  The number of patients discontinuing treatment due to adverse events will be assessed between low dose treatment, high dose treatment, and placebo groups
Change in transcriptomic profile from baseline, as measured by RNA-seq (transcriptome biomarker analysis) | 20 weeks
  Transcriptome biomarker analysis is widely used to assess dynamic changes in biological systems in response to disease processes and applied stimuli, which cannot be captured with genomic sequencing of DNA mutations and variations. Unravel Biosciences has created a proprietary algorithm for analyzing transcriptome data, identifying underlying signatures of disease progression or recovery. The machine learned gene network approach predicted the use of vorinostat based on restoring a transcriptome signature of Rett syndrome toward a healthy state, which was confirmed preclinically and motivated this clinical trial. The same algorithm will be used to assess time-dependent changes in the transcriptome network signature, to evaluate its ability to capture clinical response data and to measure the extent of restoration of a disease signature back to a healthy state in a human relative to pre-clinical models.

SECONDARY OUTCOMES:
Change from baseline on PTHS-specific Clinical Global Impression Improvement Scale (CGI-I) | 20 weeks
  7 point Likert scale with 1=very much improved and 7=very much worse
Change from baseline in PTHS-specific Clinical Global Impression Severity Scale (CGI-S) | 20 weeks
  7 point Likert Scale; 1=normal, 7=extremely ill
Change from baseline in the Caregiver Impression of Improvement scale (CareGI-I) | 20 weeks
  A 5-point Likert scale is used with the following response options: Much Improved (1); Improved (2); Unchanged (3); Worse (4); or Much Worse (5).
Change from baseline in the Revised Motor Behavioral Assessment (R-MBA) | 20 weeks
  Each of the 24 assessment items are scored based on observed or recently reported severity/frequency and scored on a five-point Likert scale between 0 and 4, with higher numbers denoting higher levels of severity/frequency.
Change from baseline in Observer-Reported Communication Ability Measure (ORCA) | 20 weeks
  The ORCA measure consists of 84 total questions with 70 behavioral items within 22 concepts/functions (e.g., refuse object, make choices) that cover expressive, receptive and pragmatic areas of communication, alongside a set of 14 descriptive items that capture important information about the individual's unique ways of communicating. The questionnaire is designed to be completed by the primary caregiver who is most familiar with the individual and the ways they communicate. ORCA measure scoring is done by dedicated statistical algorithm provided by Duke University and response items are not measured using a simple numerical rating scale.
Change from baseline in the International Cooperative Ataxia Rating Scale (ICARS) | 20 weeks
  A total of 19 questions with four subscale domains is used for assessment. Total possible score = 100, with lower scores representing lower disease burden.
Changes in sleeping habits as measured by modified Child Sleep Habits Questionnaire (CSHQ) | 20 weeks
  A modified version of the 45-item caregiver questionnaire will be used. Items are rated on a three-point scale: "usually" if the sleep behavior occurred five to seven times/week; "sometimes" for two to four times/week; and "rarely" for zero to one time/week. Lower scores are suggestive of lower disease burden on sleep behavior
Change in revised Face Legs Activity Cry and Consolability (FLACC) observational pain tool | 20 weeks
  The Face Legs Activity Cry and Consolability (FLACC) tool is a behavioral pain assessment scale used for nonverbal patients who are unable to self-report their level of pain. Pain is assessed through observation of 5 categories including face, legs, activity, cry, and consolability. Each category is scored from 0 to 2 to provide a total score ranging from 0 to 10. Higher scores represent greater symptom burden. The revised FLACC (Malvya, et.al., 2006) incorporates pain behaviors more often observed in cognitively impaired adults and children and has been demonstrated to have a reasonable level of reliability and validity for use in assessing pain in nonverbal children with cognitive impairment.
Reduction in seizure frequency as measured by seizure diary | 20 weeks
  Caregiver-recorded seizure frequency, duration, and quality will be evaluated for evidence of improvement based on reduction in seizure burden
GI symptom measures relative to baseline using a subset of questions from the Gastrointestinal Symptom Rating Scale (GSRS) | 20 weeks
  A subset of 7 questions from the GSRS will be used in the study, each question rated on a 4 point ordinal scale, "0" representing no symptoms and "3" representing significant symptom burden. Lower scores reflect lower symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Neal I Muni, M.D., MSPH, Study Director — Unravel Biosciences, Inc.
Locations (1):
- Grupo de Investigación Clínica PECET (GIC-PECET), Medellín, Colombia

IPD SHARING:
Plan to Share IPD: No